CLINICAL TRIAL: NCT03456973
Title: Nurse AMIE: A Tablet Based Supportive Care Platform in Metastatic Breast Cancer (AMIE = Addressing Metastatic Individuals Everyday)
Brief Title: Nurse AMIE: A Tablet Based Supportive Care Platform in Metastatic Breast Cancer
Acronym: NurseAMIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006544
Record Dates: First submitted 2017-06-06; First posted 2018-03-07 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse AMIE (Experimental)
  Interventions: Behavioral: Nurse AMIE

INTERVENTIONS:
Behavioral: Nurse AMIE — Supportive care software platform

SUMMARY:
The investigators propose to build and test a supportive care software platform called Nurse AMIE (Addressing Metastatic Individuals Everyday) to be provided to metastatic breast cancer patients on Android Tablets. This program will be tested in 50 metastatic breast cancer patients within the Penn State Cancer Institute's 28 county catchment area. The company with whom the investigator will partner to develop this application is already working with multiple investigators at the institution (Webster Group).

DETAILED DESCRIPTION:
Goals of the Nurse AMIE software program are to regularly assess psychosocial, functional, and symptom needs among metastatic breast cancer patients and to provide appropriate interventions via YouTube style videos, weekly Skype calls (face to face, tablet to tablet) with a patient navigator at Penn State, and appropriate referrals to phone or in person consultations as needed. The proposed Nurse AMIE software program will allow for the provision of resources (YouTube style videos, audio files, exercises) to intervene on many of the common symptoms and challenges experienced by metastatic patients. This is an identified need on the part of both metastatic patients and their medical care teams. Finally, it will also allow patient navigators to check in with patients, reviewing responses to surveys, discerning whether new or different interventions are needed, and connecting women to palliative care and other services if additional care is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Women with metastatic breast cancer
2. ECOG performance score ≤3.
3. English Speaking
4. With sufficient vision/hearing or family support

Exclusion Criteria:

1. Medical or psychiatric conditions (beyond breast cancer, its treatment, and its symptoms) that would impair our ability to test study hypotheses (e. g. psychotic disorders, dementia, inability to give informed consent or follow the instruction).
2. Patients who are receiving any other behavioral intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Feasibility- the proportion of patients who interact at least one month with tablet. | 3 months
  The proportion of women who consent, take a tablet home, who actually interact with the tablet and participate at least one month of the program.

SECONDARY OUTCOMES:
Acceptability - the proportion of patients who agree to participate | 3 months
  The proportion of patients who agree to participate among those deemed eligible and cleared by oncologist.

OTHER OUTCOMES:
Examine the effects of the program on quality of life | 3 months
  This will be compared using surveys at the beginning and end of the study period (3 months)
Qualitative assessment of physician, patient, and navigator endorsement of the program. | 1 month.
  At the conclusion of the study, physicians, patients and navigators will be asked semi-structured qualitative questions
Physical Function: Short Physical Performance Battery | 9 months
  Objectively-measured physical function will be assessed using the Short Physical Performance Battery (SPPB).
  The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn H Schmitz, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oostra DL, Burse NR, Wolf LJ, Schleicher E, Mama SK, Bluethmann S, Schmitz K, Winkels RM. Understanding Nutritional Problems of Metastatic Breast Cancer Patients: Opportunities for Supportive Care Through eHealth. Cancer Nurs. 2021 Mar-Apr 01;44(2):154-162. doi: 10.1097/NCC.0000000000000788. PMID 32022781